CLINICAL TRIAL: NCT01417351
Title: Assessment of Inflammatory Markers and Pregnancy Outcomes in Vitamin D-Supplemented Women at Risk of Vitamin D Deficiency: A Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Vitamin D Supplementation During Pregnancy on Clinical Outcomes and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 217516
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Vitamin D Deficiency
Keywords: pregnancy; immune function
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 400 IU Vitamin D3 (Placebo Comparator): Women in this study arm receive 400 IU of vitamin D3 per day, or what is in a standard prenatal multivitamin. They also receive a placebo study supplement.
  Interventions: Dietary Supplement: 400 IU vitamin D3
- 2,000 IU Vitamin D3 (Experimental): Women in this arm receive 2,000 IU vitamin D per day: 400 IU from a standard prenatal multivitamin plus an additional 1,600 IU vitamin D3 in the study supplement.
  Interventions: Dietary Supplement: 2,000 IU Vitamin D3

INTERVENTIONS:
Dietary Supplement: 400 IU vitamin D3 — Women in this study arm receive 400 IU of vitamin D3 per day, or what is in a standard prenatal multivitamin. They also receive a placebo study supplement.
  Arms: 400 IU Vitamin D3
Dietary Supplement: 2,000 IU Vitamin D3 — Women in this arm receive 2,000 IU vitamin D per day: 400 IU from a standard prenatal multivitamin plus an additional 1,600 IU vitamin D3 in the study supplement.
  Arms: 2,000 IU Vitamin D3

SUMMARY:
Researchers at the USDA Western Human Nutrition Research Center and clinicians at UC Davis Medical Center are currently conducting a study on the effects of vitamin D supplementation during pregnancy on maternal health and immune function. The investigators believe that vitamin D supplementation at levels greater than the current recommendation is beneficial for maternal health during pregnancy. In particular, there is evidence that vitamin D deficiency during pregnancy puts women at greater risk for diseases like pre-eclampsia, which may be due to an imbalance in immune function at the placenta. This randomized, double-blind study is designed to test this hypothesis. Pregnant women who participate in the study receive either 400 IU or 2,000 IU of vitamin D per day for the duration of their pregnancy. The investigators will collect blood at three time points during pregnancy (16-20 weeks, 26-28 weeks, 36 weeks gestation) for analysis of immune function and vitamin D status. The investigators are also collecting data on clinical parameters, such as blood pressure and glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Less than 20 weeks gestation
* Over 18 years of age
* Able to swallow nutritional supplements

Exclusion Criteria:

* Use of medications known to affect vitamin D metabolism
* Diagnosis of type 1 diabetes
* History of thyroid, renal, or liver disease
* Problems with digestion or absorption

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in T-cell cytokine expression | 16-20 wks, 26-28 wks, and 36 wks gestation
  Inflammatory and regulatory cytokines will be measured in cultured T-cells by flow cytometry.

SECONDARY OUTCOMES:
Change in Vitamin D status | 16-20 wks, 26-28 wks, 36 wks gestation
  Serum 25-OH vitamin D and 1, 25 (OH)2 Vitamin D
Change in innate immune function | 16-20 wks, 26-28 wks, 36 wks gestation
  Monocyte and NK cell cytokine expression and response to stimulation with Toll-like Receptor agonists.
Change in blood pressure | 16-20 wks, 26-28 wks, 36 wks gestation
  Blood pressure will be measured using standard techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Stephensen, PhD, Study Director — USDA, ARS, Western Human Nutrition Research Center
Locations (2):
- United States (2):
  - USDA-Western Human Nutrition Research Center, Davis, California
  - UC Davis Medical Center Obstetrics & Gynecology, Sacramento, California

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Zerofsky MS, Jacoby BN, Pedersen TL, Stephensen CB. Daily Cholecalciferol Supplementation during Pregnancy Alters Markers of Regulatory Immunity, Inflammation, and Clinical Outcomes in a Randomized Controlled Trial. J Nutr. 2016 Nov;146(11):2388-2397. doi: 10.3945/jn.116.231480. Epub 2016 Sep 21. PMID 27655755